CLINICAL TRIAL: NCT06304636
Title: Descartes-15 for Patients With Relapsed/Refractory Multiple Myeloma
Acronym: DC15-MM-01
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Phase 1 enrollment completed. Further clinical development terminated
Sponsor: Cartesian Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DC15-MM-01
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Refractory Multiple Myeloma; Relapsed Multiple Myeloma
Keywords: Relapsed/Refractory; Relapsed Myeloma; Refractory Myeloma; Multiple Myeloma; Car-T; CART; Descartes-15; Descartes; Myeloma; T cells; cell gene
MeSH Terms: conditions — Multiple Myeloma; Recurrence; Neoplasms, Plasma Cell

STUDY DESIGN:
Intervention Model Description: Study consists of two parts. Part 1 is a single-arm dose escalation study. Part 2 is a dose-expansion study with 2 arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Descartes-15 with lymphodepletion (Experimental): Intra-patient dose escalation arm with three dose levels over the course of six infusions of cell product. Patients will receive lymphodepletion prior to initiating cell therapy.
  Interventions: Drug: Descartes-15
- Part 2 Arm 1 Descartes-15 with lymphodepletion (Experimental): Descartes-15 infusions at the maximum tolerated dose level from Part 1. Patients will receive lymphodepletion prior to initiating cell therapy.
  Interventions: Drug: Descartes-15
- Part 2 Arm 2 Descartes-15 without lymphodepletion (Experimental): Descartes-15 infusions at the maximum tolerated dose level from Part 1. Patients will not receive lymphodepletion prior to initiating cell therapy.
  Interventions: Drug: Descartes-15

INTERVENTIONS:
Drug: Descartes-15 — Autogolous T-cells expressing a chimeric antigen receptor directed to BCMA

SUMMARY:
This is a Phase I dose-escalation study to evaluate the safety, tolerability and preliminary efficacy of an autologous BCMA-targeting RNA-engineered CAR T-cell therapy in patients with Relapsed/Refractory Multiple Myeloma. The cell product is referred to as Descartes-15

ELIGIBILITY:
Inclusion Criteria

* Patients must be 18 years of age or older at the time of enrollment.
* Patients must be diagnosed with active and measurable relapsed/refractory multiple myeloma.
* Patients must have failed at least 3 prior lines of therapy which must have included an immunomodulatory drug, a proteasome inhibitor, and an anti-CD38 drug or biologic. Failure of treatment and measurable myeloma disease are defined as per 2016 IMWG criteria.
* Patients must have clinical performance status of ECOG 0-2.
* Patients must have adequate vital organ function as defined by:
* Hemoglobin ≥8 g/dL
* Absolute neutrophil count > 1000/ mm3
* Platelets > 50,000/mm3
* ALT/AST levels lower than 3-fold of normal
* Creatinine clearance ≥45 mL/min/1.73 m2
* Normal cardiac and pulmonary function
* No thromboembolic events in the past 3 months
* No heparin allergy or active infection

Exclusion Criteria

* Patients who have any active and uncontrolled infection.
* Ongoing treatment with chronic immunosuppressants (e.g., cyclosporine or systemic steroids above 40 mg/day prednisone equivalent).
* Patients who have active central nervous system disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Determine the safety of Descartes-15 in patients with relapsed/refractory multiple myeloma (R/R MM) | Day -60 to Month 12
  Results will be descriptive. Safety and tolerability endpoints are adverse events and serious adverse events as proportion of all participants at a given dose level and in the overall study population.

SECONDARY OUTCOMES:
To assess the anti-myeloma activity of Descartes-15, as measured by IMWG response criteria and progression-free survival | Day 1 to Month 12
  Efficacy will be assessed by descriptive statistics of treatment response per IMWG criteria. Efficacy endpoints will be reported as proportion of participants achieving Stable Disease (SD), Partial Response (PR), Very Good Partial Response (VGPR), Complete Response (CR) and stringent Complete Response (sCR) as the best response at a given dose level and in the overall study population.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Cancer and Blood Disorders (AON), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No